CLINICAL TRIAL: NCT01905540
Title: A Phase 1, Open-label, Randomized, 3-Period, Relative Bioavailability Study Comparing the Pharmacokinetics of SSP-004184AQ (Magnesium Salt) to SSP-004184SS (Disodium Salt) Each Administered as a Single Dose and as Two Doses of SSP-004184 (Free Acid) in Healthy Adult Subjects
Brief Title: A Relative Bioavailability Study of SSP-004184AQ (Magnesium Salt) and SSP-004184SS (Disodium Salt)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SPD602-111
Record Dates: First submitted 2013-07-18; First posted 2013-07-23 (Estimated); Results first posted 2014-12-24 (Estimated); Last update posted 2021-07-19 (Actual); Status verified 2021-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- SSP-004184AQ (single dose) (Experimental): 40 mg/kg (oral capsule form) given once on Day 1
  Interventions: Drug: SSP-004184AQ
- SSP-004184SS (single dose) (Experimental): 21.8 mg/kg (oral capsule form) given once on Day 1
  Interventions: Drug: SSP-004184SS
- SSP-004184AQ (2 doses) (Experimental): 40 mg/kg (oral capsule form) given twice (12 hours apart) on Day 1
  Interventions: Drug: SSP-004184AQ
- SSP-004184SS (2 doses) (Experimental): 21.8 mg/kg (oral capsule form) given twice (12 hours apart) on Day 1
  Interventions: Drug: SSP-004184SS

INTERVENTIONS:
Drug: SSP-004184AQ — Magnesium salt
  Other Names: SPD602
  Arms: SSP-004184AQ (2 doses); SSP-004184AQ (single dose)
Drug: SSP-004184SS — Disodium salt
  Other Names: SPD602
  Arms: SSP-004184SS (2 doses); SSP-004184SS (single dose)

SUMMARY:
This study will evaluate the relative bioavailability of the new SSP-004184SS capsule formulation compared to the original SSP-004184AQ drug plus excipients formulation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Must be considered "healthy".
* Serum ferritin >20ng/mL, hemoglobin >125g/L and erythrocyte indices within normal range

Exclusion Criteria:

* Subject has a clinically significant history or a disorder detected during the medical interview/physical examination at the Screening Visit or any other medical condition that is capable of altering the absorption, metabolism, or elimination of drugs
* Acute illness, as judged by the investigator, within 2 weeks of Day 1 of Treatment Period 1.
* Known or suspected intolerance or hypersensitivity to the investigational products, closely related compounds, or any of the stated ingredients.
* Subject has a history of thyroid disorder that has not been stabilized on thyroid medication or treatment within 3 months
* History of alcohol or other substance abuse within the last year.
* A positive screen for alcohol or drugs of abuse at the Screening Visit.
* Confirmed systolic blood pressure >139mmHg or <89mmHg, and diastolic blood pressure >89mmHg or <49mmHg.
* Twelve-lead ECG demonstrating QTc >450msec at screening.
* Routine consumption of more than 2 units of caffeine per day or subjects who experience caffeine withdrawal headaches.
* Male subjects who consume more than 3 units of alcohol per day. Female subjects who consume more than 2 units of alcohol per day.
* A positive HIV antibody screen, HBsAg, or HCV antibody screen.
* Use of tobacco in any form (eg, smoking or chewing) or other nicotine-containing products in any form (eg, gum, patch) within 30 days prior to Day 1 of Treatment Period 1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-08-05 (Actual); Primary Completion 2013-09-20 (Actual); Study Completion 2013-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Clinical Pharmacology of Miami, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- AQ-SS-AQ2: SSP-004184AQ 40mg/kg as a single dose, followed by SSP-004184SS 21.8mg/kg as a single dose, followed by SSP-004184AQ 40mg/kg as a morning and evening dose.
- AQ-SS-SS2: SSP-004184AQ 40mg/kg as a single dose, followed by SSP-004184SS 21.8mg/kg as a single dose, followed by SSP-004184SS 21.8mg/kg as a morning and evening dose.
- SS-AQ-AQ2: SSP-004184SS 21.8mg/kg as a single dose, followed by SSP-004184AQ 40mg/kg as a single dose, followed by SSP-004184AQ 40mg/kg as a morning and evening dose.
- SS-AQ-SS2: SSP-004184SS 21.8mg/kg as a single dose, followed by SSP-004184AQ 40mg/kg as a single dose, followed by SSP-004184SS 21.8mg/kg as a morning and evening dose.
Period: Period 1
Arm/Group | AQ-SS-AQ2 | AQ-SS-SS2 | SS-AQ-AQ2 | SS-AQ-SS2
Started | 7 | 7 | 7 | 7
Completed | 7 | 7 | 7 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | AQ-SS-AQ2 | AQ-SS-SS2 | SS-AQ-AQ2 | SS-AQ-SS2
Started | 7 | 7 | 7 | 7
Completed | 7 | 7 | 7 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | AQ-SS-AQ2 | AQ-SS-SS2 | SS-AQ-AQ2 | SS-AQ-SS2
Started | 7 | 7 | 7 | 7
Completed | 6 | 7 | 6 | 6
Not Completed | 1 | 0 | 1 | 1
Not completed — Other | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Set: All enrolled subjects who had taken at least 1 dose of investigational product and had at least 1 post-dose safety assessment (defined as treatment emergent adverse events [TEAEs], physical examination findings, clinical laboratory test results, vital sign measurements, and 12-lead ECG readings).
Groups:
- Total: Total of all reporting groups
Arm/Group | AQ-SS-AQ2 | AQ-SS-SS2 | SS-AQ-AQ2 | SS-AQ-SS2 | Total
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.7 (12.58) | 44.4 (11.53) | 41.3 (10.27) | 42.7 (13.46) | 43 (11.4)
Age, Customized [Count of Participants; unit: Participants]
  >=65 years | 1 | 0 | 0 | 0 | 1
  Between 18 and 65 years | 6 | 7 | 7 | 7 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 2 | 7
  Male | 5 | 5 | 6 | 5 | 21
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 7 | 7 | 7 | 7 | 28

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Steady-state Plasma Concentration-time Curve (AUClast) of SSP-004184 After One Dose
Description: AUC 0-last is the area under the plasma concentration versus time curve from time 0 to the time of last quantifiable concentration. AUC can be used as a measure of drug exposure. It is derived from drug concentration and time so it gives a measure how much and how long a drug stays in a body
Time Frame: Periods 1 & 2: Within 30 min pre-dose, and Post-dose 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 24, 48, 72, 96, and 120 hrs. Period 3: Within 30 min pre-dose, and Post-dose 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 12.5, 13, 13.5, 14, 14.5, 16, 20, 24, 48, 72, 96, and 120 hrs.
Population: Pharmacokinetic Set: All subjects who had taken at least 1 dose of investigational product, had at least 1 post-dose safety assessment, and for whom the primary pharmacokinetic data were considered sufficient and interpretable.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | SSP-004184AQ (Single Dose) | SSP-004184SS (Single Dose)
Number analyzed (Participants) | 28 | 28
ng*h/mL | 261901.9 (71252.3) | 164340 (43914)
Statistical Analysis 1: Comparison: SSP-004184AQ (Single Dose) vs SSP-004184SS (Single Dose); Test type: Non-Inferiority or Equivalence — The statistical comparison of log-transformed pharmacokinetic parameters between the single-dose treatment groups (Treatments AQ and SS) was based on the 90% CI for the ratio of the geometric means. If the 90% CI was entirely contained within the acceptance range of 0.8-1.25 then it was concluded that there was no statistically significant difference between treatments for the relevant parameter. Doses were normalized to the SSP-004184AQ (40mg/kg) dose prior to statistical analysis; Ratio of geometric LS means = 1.244, 90% CI 2-sided [1.081 to 1.430]

2. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC) From Time Zero to Infinity (AUCinf) of SSP-004184 After One Dose
Description: AUCinf is the area under the curve extrapolated to infinity, calculated using the observed value of the last nonzero concentration. AUC can be used as a measure of drug exposure. It is derived from drug concentration and time so it gives a measure how much and how long a drug stays in a body.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | SSP-004184AQ (Single Dose) | SSP-004184SS (Single Dose)
Number analyzed (Participants) | 26 | 28
ng*h/mL | 263911.3 (68979.4) | 164614.8 (43858.8)
Statistical Analysis 1: Comparison: SSP-004184AQ (Single Dose) vs SSP-004184SS (Single Dose); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric LS Means = 1.233, 90% CI 2-sided [1.070 to 1.422]

3. Primary Outcome: Maximum Plasma Concentration (Cmax) of SSP-004184 After One Dose
Description: Cmax is a term that refers to the maximum (or peak) concentration that a drug achieves in the body after the drug has been administrated
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SSP-004184AQ (Single Dose) | SSP-004184SS (Single Dose)
Number analyzed (Participants) | 28 | 28
ng/mL | 110114.3 (26503) | 77068.6 (21198.9)
Statistical Analysis 1: Comparison: SSP-004184AQ (Single Dose) vs SSP-004184SS (Single Dose); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric LS means = 1.344, 90% CI 2-sided [1.135 to 1.592]

4. Secondary Outcome: Area Under the Steady-state Plasma Concentration-time Curve (AUClast) of SSP-004184 After Two Doses
Description: AUClast is the area under the concentration versus time curve from the time of dosing to the last measurable concentration. AUC can be used as a measure of drug exposure. It is derived from drug concentration and time so it gives a measure how much and how long a drug stays in a body.
Time Frame: as for outcome 1
Population: Pharmacokinetic Set: All subjects who had taken at least 1 dose of investigational product and had at least 1 post-dose safety assessment and for whom the primary pharmacokinetic data were considered sufficient and interpretable.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- SSP-004184AQ (2 Doses): SSP-004184AQ 40mg/kg morning and evening dose.
- SSP-004184SS (2 Doses): SSP-004184SS 21.8mg/kg morning and evening dose
Arm/Group | SSP-004184AQ (2 Doses) | SSP-004184SS (2 Doses)
Number analyzed (Participants) | 12 | 13
ng*hr/mL | 545957 (186707.3) | 294186.8 (78102.1)

5. Secondary Outcome: Area Under the Plasma Concentration-time Curve (AUC) From Time Zero to Infinity (AUCinf) of SSP-004184 After Two Doses
Description: AUCinf is the area under the plasma concentration versus time curve extrapolated to infinity, calculated using the observed value of the last nonzero concentration. AUC can be used as a measure of drug exposure. It is derived from drug concentration and time so it gives a measure how much and how long a drug stays in a body.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | SSP-004184AQ (2 Doses) | SSP-004184SS (2 Doses)
Number analyzed (Participants) | 12 | 10
ng*hr/mL | 546114.1 (186698.2) | 294758.5 (81194.7)

6. Secondary Outcome: Maximum Plasma Concentration (Cmax) of SSP-004184 After Two Doses
Description: as for outcome 3
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SSP-004184AQ (2 Doses) | SSP-004184SS (2 Doses)
Number analyzed (Participants) | 12 | 13
ng/mL
  Dose 1 | 112558.3 (28036.8) | 77958.3 (34372.5)
  Dose 2 | 73776.9 (17193.2) | 43015.4 (11168.8)

ADVERSE EVENTS:
Description: The Safety Set was defined as all enrolled subjects who had taken at least 1 dose of investigational product and had at least 1 post-dose safety assessment (defined as treatment emergent adverse events (TEAEs), physical examination findings, clinical laboratory test results, vital sign measurements, and 12-lead ECG readings).
Groups:
- SSP-004184AQ (Single Dose): SSP-004184AQ: 40mg/kg (equivalent to 36.2mg/kg free-acid dose) administered as a single dose in a fasted state in the morning.
- SSP-004184SS (Single Dose): SSP-004184SS: 21.8mg/kg (equivalent to 18.1mg/kg free-acid dose) administered as a single dose in a fasted state in the morning.
- SSP-004184AQ (2 Doses): SP-004184AQ: 40mg/kg (equivalent to 36.2mg/kg free-acid dose) administered in the morning and 40mg/kg administered 12 hours later.
- SSP-004184SS (2 Doses): SSP-004184SS: 21.8mg/kg (equivalent to 18.1mg/kg free-acid dose) administered in the morning and 21.8mg/kg administered 12 hours later.
Arm/Group | SSP-004184AQ (Single Dose) | SSP-004184SS (Single Dose) | SSP-004184AQ (2 Doses) | SSP-004184SS (2 Doses)
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 12/28 | 11/28 | 5/12 | 5/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SSP-004184AQ (Single Dose) (N=28) | SSP-004184SS (Single Dose) (N=28) | SSP-004184AQ (2 Doses) (N=12) | SSP-004184SS (2 Doses) (N=13)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 2 (2) | 0 (0) | 2 (2)
Chromaturia (Renal and urinary disorders) | 12 (12) | 9 (9) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.